CLINICAL TRIAL: NCT06974773
Title: At-Home Transcranial Direct Current Stimulation (tDCS) Using the NettleEndo Device for Reducing Symptoms of Endometriosis - A Pivotal Double-Blind, Randomized, Placebo-Controlled Clinical Trial
Brief Title: Remote Electrical Stimulation as a Long-term Intervention for Endometriosis Flare Ups
Acronym: RELIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samphire Group, Inc. (Industry)
Collaborators: Alethios, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RELIEF25
Record Dates: First submitted 2025-05-06; First posted 2025-05-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
Keywords: Endometriosis; Dysmenorrhea; Chronic Pelvic Pain; tDCS; Neuromodulation; Women's Health
MeSH Terms: conditions — Endometriosis; Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel assignment clinical trial in which participants are randomly assigned in a 1:1 ratio to receive either active transcranial direct current stimulation (tDCS) or sham stimulation using the NettleEndo wearable device. Each participant remains in their assigned group throughout the 12-week intervention period. The study is double-blind: neither participants nor outcome assessors know group assignment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS - NettleEndo Device (Experimental): Participants assigned to this arm will receive active transcranial direct current stimulation (tDCS) using the NettleEndo wearable device. The device delivers 2 mA of stimulation for 20 minutes per session, five sessions per week, for a total of 12 weeks. Stimulation is delivered over the left primary motor cortex (M1) and dorsolateral prefrontal cortex (DLPFC) using pre-programmed settings. Participants complete all sessions at home and log outcomes via a mobile app. Device use is monitored remotely through digital logs.
  Interventions: Device: NettleEndo
- Sham tDCS - NettleEndo Device (Sham Comparator): Participants assigned to this arm will receive sham transcranial direct current stimulation (tDCS) using the NettleEndo wearable device. The device mimics the sensation of active stimulation by ramping up to 2 mA for 20 seconds before turning off, with no therapeutic current delivered for the remainder of the 20-minute session. Participants use the device five times per week for 12 weeks. Sessions are completed at home, and outcome measures are recorded via a mobile app. Device use is remotely monitored via app-based logging. Participants and investigators are blinded to group allocation.
  Interventions: Device: Sham NettleEndo Device

INTERVENTIONS:
Device: NettleEndo — The NettleEndo device is a portable, home-use transcranial direct current stimulation (tDCS) system designed to deliver low-intensity electrical stimulation to targeted brain regions. The device delivers a constant current of 2 mA in the active stimulation group, targeting the left primary motor cortex (M1) and left dorsolateral prefrontal cortex (DLPFC) through pre-set electrode positioning.
  Arms: Active tDCS - NettleEndo Device
Device: Sham NettleEndo Device — The sham version of the NettleEndo device is visually identical to the active device and is used under the same schedule. The device is pre-programmed to deliver a brief 2 mA current for 20 seconds at the beginning of each session to mimic the initial skin sensations of active stimulation, after which no current is delivered for the remainder of the session. This allows participants to remain blinded to their group assignment. The device is used with the same electrode positioning as the active version.
  Arms: Sham tDCS - NettleEndo Device

SUMMARY:
The goal of this clinical trial is to learn if a wearable brain stimulation device called NettleEndo can reduce chronic pelvic pain and improve wellbeing in women with endometriosis. The study also aims to assess the safety and usability of the device when used at home over several months.

The main questions it aims to answer are:

1. Does at-home transcranial direct current stimulation (tDCS) reduce daily pain intensity in women with endometriosis?
2. Does the device also improve mood and sleep quality?

Researchers will compare two groups-one receiving active brain stimulation and one receiving a sham (placebo) stimulation-to see if the active device provides greater improvements in symptoms.

Participants will:

1. Use the NettleEndo device at home for 20 minutes per session, five times per week for 12 weeks
2. Be randomly assigned to receive either real or sham stimulation through the device
3. Complete daily and weekly symptom ratings through a mobile app
4. Be followed for 90 days after completing the intervention to monitor longer-term effects

All activities are completed remotely using a smartphone app. Participants can contact the study team with questions at any time. The study is double-blind, meaning neither participants nor the researchers assessing outcomes will know who received active or sham treatment until the end of the trial.

DETAILED DESCRIPTION:
This is a decentralized, randomized, double-blind, sham-controlled clinical trial evaluating the efficacy, safety, and usability of the NettleEndo device for managing endometriosis-associated symptoms. The device delivers transcranial direct current stimulation (tDCS) and is used at home for 20 minutes per session, five sessions per week, over 12 weeks. The stimulation targets the left dorsolateral prefrontal cortex (DLPFC) and primary motor cortex (M1), both of which are involved in the modulation of pain and emotional regulation.

Participants are randomly assigned in a 1:1 ratio to receive either active or sham stimulation. The sham group receives a brief stimulation ramp-up (2 mA for 20 seconds) to mimic sensation but no sustained current. All participants use the same wearable device, complete self-report measures through a mobile app, and are blinded to group assignment.

Data are collected using the Alethios platform, a compliant digital health system that supports electronic informed consent, daily and monthly questionnaires, adverse event tracking, and automated session logging. Optional wearable integration allows for passive data capture, including sleep, activity, and heart rate variability.

The trial includes a 12-week treatment period followed by a 90-day follow-up phase. Outcomes include pain intensity, mood, sleep, and quality of life. Randomization is stratified by pain level and menstrual cycle status. Interim analyses are planned after approximately one-third and two-thirds of participants complete the intervention.

ELIGIBILITY:
Inclusion Criteria

* Female, 22-45 years old
* Assigned female at birth
* Fluent in English
* Capacity to consent
* Confirmed diagnosis of endometriosis by a qualified physician, via:
* Laparoscopic surgery with biopsy-proven endometriosis, OR
* Clear evidence of ovarian endometrioma or deep infiltrating endometriosis on ultrasound/MRI
* Pain levels:

For menstruating participants, all of the following need to be met:

* Regular menstrual cycles (21-35 days)
* Mean DYS NRS ≥4 during menstrual bleeding days (over the last 28 days, self-assessed)
* AND Mean NMPP NRS ≥4 during non-menstrual days (over the last 28 days, self-assessed)

For non-menstruating patients, all required:

* Irregular/absent cycles OR post-hysterectomy OR surgically menopausal
* Mean pelvic pain NRS ≥4 (over the last 28 days, self-assessed)
* Pain present on ≥50% of days
* Access to a smartphone with an internet data plan, phone must be iOS 13.4+, or Android 12+.
* No hormonal contraception or at least 6 months of consistent adherence to any hormonal contraception (e.g., IUD, pill, injection).
* Capacity to follow instructions and operate the study device.

Exclusion Criteria

* Pregnancy/breastfeeding or planning to become pregnant in next 6 months
* History of epileptic neurological conditions in the immediate family
* Severe/untreated neurological disease (e.g., epilepsy or seizure disorders, stroke or transient ischemic attack [TIA], subarachnoid hemorrhage, traumatic brain injury [TBI] with persistent neurological deficits, brain tumors [malignant or benign], multiple sclerosis, Parkinson's disease, Alzheimer's disease or other dementias, Huntington's disease, cerebral aneurysms or arteriovenous malformations [AVMs], active central nervous system infections [e.g., meningitis, encephalitis], hydrocephalus, other neurodegenerative diseases not otherwise specified, or any other neurological condition that, in the opinion of the principal investigator, may increase risk or interfere with study participation or outcomes)
* Metal implants/electronic devices in brain, head, or neck area
* Participating in any other clinical trial
* History of stroke, brain surgery, tumors, head trauma
* Active skin lesions, open wounds, cuts, or infections on the scalp
* Active scalp conditions (dermatitis, eczema, psoriasis)
* Significant scarring/burns/other skin damage on scalp
* Schizophrenia or bipolar disorder
* History of suicidal behavior or clinically significant self-injurious behavior (e.g., one or more suicide attempts, non-suicidal self-injury [NSSI], or other behaviors indicative of intent to harm oneself), as determined by participant self-report.
* Treatment plan must be stabilized (≥6 weeks analgesic/ ≥6 months hormonal contraception, and crucially no new medication changes before randomization)
* Planning to commence any new treatment during intervention period
* Lack of capacity to consent
* Participation in a neurotechnology or drug trial in the last 6 months.
* Recent surgical intervention for endometriosis within 6 months of enrollment or planned surgical intervention for endometriosis during the study period.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in daily endometriosis-associated pain intensity (NRS) | Daily, throughout the study (6 months)
  Average change from baseline in daily self-reported pain intensity related to endometriosis, using a 0-10 Numerical Rating Scale (NRS). This will be measured separately for dysmenorrhea (Dysmenorrhea NRS; DYS NRS) and non-menstrual pelvic pain (Non-Menstrual Pelvic Pain; NMPP NRS). Collected via mobile app. A decrease in NRS, NMPP NRS and DYS NRS scores indicate a better outcome, as it reflects reduced pain intensity.

SECONDARY OUTCOMES:
Change in endometriosis-specific quality of life (EHP-30) | Monthly starting at baseline until the end of the study (6 months)
  Change from baseline in total and subscale scores on the Endometriosis Health Profile-30 (EHP-30), a 30-item scale assessing the quality of life specific to endometriosis. Each item is rated on a 5-point Likert scale (1 = "Not at all," 5 = "Extremely"). The scale includes subscales for Pain, Work, Social Relationships, Health, Sexual Activity, and Emotion, each with its own set of items. The total score ranges from 0 to 120, where 0 = No impact on quality of life and 120 = Maximum impact on quality of life. A higher score indicates worse quality of life.
Change in general health status (EQ-5D-5L) | Monthly starting at baseline until the end of the study (6 months)
  Change from baseline in EQ-5D-5L index scores, a 5-item scale assessing general health status. Each item is rated on a 5-point Likert scale (1 = No problems, 5 = Unable to do). The total index score is calculated based on responses across all five domains, with the score ranging from 0 (representing worst possible health) to 1 (representing best possible health). A higher score indicates better health status.
Change in severity of illness and improvement over time (CGI) | Monthly starting at baseline until the end of the study (6 months)
  The Clinical Global Impressions (CGI) scale is a brief, 3-item rating tool used by clinicians to assess the severity of a patient's illness, their improvement over time, and the efficacy of their treatment.

OTHER OUTCOMES:
Device adherence (number of sessions completed) | Week 1 to Week 12
  Total number of NettleEndo sessions completed over the 12-week intervention period, recorded by the device and app logs.
Exploratory - Change in pain catastrophizing (PCS) | Monthly starting at baseline until the end of the study (6 months)
  Change from baseline in total score on the Pain Catastrophizing Scale (PCS), which consists of 13 items, each scored on a 5-point Likert scale (0 = Not at all, 4 = Extremely). The total score ranges from 0 to 52, with higher scores indicating more severe pain catastrophizing.
Exploratory - Change in insomnia severity (ISI) | Monthly starting at baseline until the end of the study (6 months)
  Change from baseline in total score on the Insomnia Severity Index (ISI), a 7-item self-report measure where each item is rated on a 0 to 4 scale. The total score is the sum of these ratings, with scores ranging from 0 to 28, where 0 = No insomnia and 28 = Severe insomnia. A higher score indicates worse insomnia severity.
Daily medication use (analgesic and hormonal) | Daily, throughout the study (6 months)
  Daily use of pain medications and hormonal treatments recorded by participants via mobile app.
Exploratory - Change in depressive symptoms (PHQ-8) | Monthly starting at baseline until the end of the study (6 months)
  Change from baseline in total score on the 8-item Patient Health Questionnaire (PHQ-8), a screening tool for depression that uses a 4-point Likert scale for each of its eight items. The total score ranges from 0 to 24, with 0 = No depressive symptoms and 24 = Severe depressive symptoms. A higher score indicates more severe depressive symptoms.
Exploratory - Change in cyclical mood and physical symptoms (DRSP) | Daily, throughout the study (6 months)
  Change in symptoms assessed using the Daily Record of Severity of Problems (DRSP), a validated tool for tracking mood, behavioural, and physical symptoms across the menstrual cycle. Participants rate symptoms daily via mobile app on a 1-6 scale, where 1 = No symptoms and 6 = Severe symptoms. A decrease in DRSP scores indicates a better outcome, reflecting reduced mood and physical symptoms.
Incidence of device-related adverse events | Week 1 to Day 90 follow-up
  Number and severity of adverse events (AEs) and serious adverse events (SAEs) deemed related to the NettleEndo device.
Menstrual cycle characteristics and timing | Daily, throughout the study (6 months)
  Participants complete daily menstruation tracking using a mobile app, recording onset and duration of bleeding.
Exploratory analysis of Heart Rate Variability (HRV) | Daily, throughout the study (6 months)
  Heart rate variability (HRV) data will be collected from participants who opt in to wearable integration. HRV will be used in exploratory analyses to assess physiological patterns during the intervention and follow-up phases.
Exploratory analysis of step count | Daily, throughout the study (6 months)
  Step count data will be collected from participants who opt in to wearable integration. Step count will be used in exploratory analyses to assess behavioural patterns during the intervention and follow-up phases.
Exploratory analysis of sleep metrics | Daily, throughout the study (6 months)
  Sleep metrics will be collected from participants who opt in to wearable integration. These data will be used in exploratory analyses to assess physiological patterns during the intervention and follow-up phases.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Shah, MD, MPH, Principal Investigator
Locations (1):
- Alethios, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No